CLINICAL TRIAL: NCT02767882
Title: Effects of Preoperative Dexamethasone in Post-operative Pain Control After Total Knee Replacement
Brief Title: Dexamethasone in Pain Control After Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW16-201
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group D1 (Active Comparator): Patients from group D will be given a bolus injection of 2 ml saline with 2 ml dexamethasone (4mg/ml) before skin incision.
  Interventions: Drug: Dexamethasone
- Group D2 (Experimental): 4ml bolus injection of dexamethasone (4mg/ml) will be given intravenously prior to incision.
  Interventions: Drug: Dexamethasone
- Group C (Placebo Comparator): 4ml bolus injection of 0.9% saline will be given intravenously prior to incision
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — Bolus injection of different dose of dexamethasone will be given intravenously prior to incision.
  Arms: Group D1; Group D2
Drug: Saline — Bolus injection of 4ml 0.9% saline will be given intravenously prior to incision.
  Arms: Group C

SUMMARY:
The primary aims of total knee replacement are improvement in functional activities and reduce pain due to degenerated knee joints. However, there are around 20-30% of patients would develop significant pain problem despite uncomplicated total knee replacement. It accounts for major post-operative problems and burdens.

Dexamethasone is glucocorticoid which is associated with anti-inflammatory response. It is well known to have prophylaxis effect for post-operative nausea and vomiting. Perioperative single dose of systemic dexamethasone have shown to be useful for reduction in pain and cumulative opioid consumption. Meta-analysis from De Oliveira et al supports that dexamethasone (up to 0.2 mg/kg) is a safe and effective multimodal pain strategy after surgical procedures. However, this dose recommendation is not surgery specific. It is essential to have more RCTs evaluating the optimal dose of steroid for pain management after hip and knee surgery.

DETAILED DESCRIPTION:
Patients will be approached at the preadmission clinic or in the general ward before operation. The analgesic methods will be explained and s/he will be recruited into the study if s/he agrees. There are standardized preoperative, intraoperative and postoperative analgesic regimes for patients undergoing total knee replacement.

For preoperative analgesic regime, pregabalin 50mg are given the night before operation. Same analgesic regime is used on the day before operation. For intraoperative regime, standardized intraarticular local anaesthetic infiltration is used. For postoperative analgesic regime, PCA using morphine is used. In addition to PCA using morphine, standardized analgesic regime is used -- regular pregabalin 50mg nocte, paracetmal 1g QID, Celebrex 200mg BD will be given for 5 days.

Patients will be randomized into one of three groups. Patients in the first group (D1) will receive standardized oral analgesic regime pre-operatively, intraoperatively and postoperatively. In addition to the above, they will be given preoperative intravenous 8mg dexamethasone. Patients in the second (D2) group will be given preoperative intravenous 16mg dexamethasone, in addition to same pre-operative, intraoperative and post-operative analgesic regimes. Patients in the third (C) group will be given preoperative intravenous 4ml 0.9% saline, in addition to same pre-operative, intraoperative and post-operative analgesic regimes.

Preoperative Care Assessment will be done at the preadmission clinic or at the general ward. Pre-operative pregabalin will be given before operation and on the day before operation. Fasting will start six hours before operation.

Range of movement of the operating knee, quadriceps function, pain scores of the affecting knee will be assessed on day before operation.

Pre-operative inflammatory marker (e.g. CRP, ESR, tumour necrosis factor α, interleukin IL-6) and H'stix will be taken on day of admission.

Anaesthetic and intraoperative care

All patients will be anaesthetized according to the following protocol:

On arrival to the operation theatre, a 18 or 16 gauge intravenous cannula will be inserted. Standard monitoring with pulse oximeter, non-invasive blood pressure, and three lead electrocardiogram will be applied prior to induction. Non-invasive blood pressure will be checked at least every 5 minutes throughout the operation.

Patients will be provided with spinal anaesthesia for the operation with 2.4 ml 0.5% heavy Marcaine will be administrated into spinal space after position confirmed with spinal needle. No intrathecal opioid will be given during the procedure. Patient will be sedated with TCI propofol (0.3 -1 ug/ml) throughout the whole total knee replacement after successful spinal anaesthesia.

Intravenous antibiotic will be given before skin incision. Hypotension will be managed with intravenous phenylephrine or ephedrine at the discretion of the anaesthesiologist. Intra-operative fluid 8-10ml/kg/hr will be infused as maintenance. Also intravenous bolus of fluid will be given for replacement of blood loss. Infusion fluid warmer and thermal blanket will be used with the aim of keeping a core temperature of 35.5-37.5 degrees Celsius.

Local anaesthetic infiltration of 40ml 0.75% ropivacaine, 0.5ml 1:200,000 adrenaline, 30mg ketorolac in 60ml normal saline will be administrated by orthopaedic surgeons after implant insertion and wound closure.

Patients will subsequently be transferred to the post anaesthetic care unit (PACU) for monitoring for at least 1 hour. H'stix and H'cue will be checked 2 hours and 4 hours after preoperative injection of dexamethasone.

Analgesic modalities and pain assessment

Procedures for the all analgesic modalities are described below:

Group D1 Patients from group D will be given a bolus injection of 2 ml saline with 2 ml dexamethasone (4mg/ml) before skin incision.

Group D2 4ml bolus injection of dexamethasone (4mg/ml) will be given intravenously prior to incision.

Group C 4ml bolus injection of 0.9% saline will be given intravenously prior to incision.

For all groups In the recovery room after surgery, boluses of 2mg intravenous morphine will be given every 5 minutes until numerical rating pain score (NRS) is less than 4/10. A PCA machine will then be connected. The machine will be configured to give 1mg of morphine at a time and the lockout duration will be set to 5 minutes. No background infusion will be given and the maximum dose limit will be 0.1mg/kg per hour of morphine sulphate.

Intramuscular morphine sulphate at a dose of 0.1mg/kg will be prescribed every 4 hours if necessary for breakthrough beginning from postoperative day 0. Intravenous 4mg ondansetron is used every 4 hours if necessary if there is any nausea or vomiting.

On postoperative day 0, patient will resume oral diet if not contraindicated. Oral paracetamol and COX-2 inhibitor will be given for 5 days. Oral pregabalin will be given for 7 days.

While on PCA morphine, the patient's respiratory rate, SpO2 and sedation score will be monitored every hour. Heart rate and blood pressure will be checked every 4 hours. NRS pain scores at rest, during knee movement, during sleep, cumulative PCA morphine doses, and number of PCA demands/goods delivered, and side effects (nausea, vomiting, dizziness) will be recorded every 4 hours. Patients will be assessed by pain team everyday.

Patients will be on PCA morphine for at least 2 days. If NRS pain scores during knee movement on postoperative day 2 is less than 4/10 or clinically low morphine consumption, PCA morphine will be stopped. PCA morphine will be continued if NRS is equal or greater than 4, or if the patient remains on a high PCA consumption.

After PCA morphine has stopped, NRS pain scores at rest and during knee movement, as well as the dose and frequency of rescue analgesia used will be charted once a day until discharge.

Surgical technique/Prosthesis The surgery will be performed by the same surgical team with standardized surgical technique. All the patients will have posterior stabilized knee prosthesis. Tranexamic acid will be given according to our protocol. Standardized regimen and technique of local infiltration of analgesic at the end of the surgery will be given as part of the multi-modal pain control protocol

Postoperative care and assessment Day zero mobilization or early mobilization with PT and OT rehabilitation is encouraged after operation. Fluid diet will be allowed on postoperative day 0.

The surgical team will assess for occurrences of postoperative surgical complications, suitability for discharge (good pain control, ambulation, normal bowel function, and ability to eat properly without vomiting. Urinary retention will be documented as well.

Range of movement of the operating knee and other rehabilitation parameters will be assessment by allied health staffs from Day 0 till day of discharge.

Side effects of steroid are documented e.g. gastrointestinal bleeding, hyperglycaemia, wound infection (Southampton wound assessment scale), or other systemic infections are documented.

Glucose level will be measured in 7am and 5pm on Day 1 and Day 2. Insulin will be used to keep glucose <15 mmol/dl. Blood investigations will also be performed. Inflammatory marker e.g. ESR, CRF, tumour necrosis factor α, interleukin IL-6 will be taken on Day 0, Day 1 and Day 2. Haemoglobin level and the need of transfusion will be documented.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80 years old
* Scheduled for elective primary unilateral total knee replacement
* Chinese patients
* Able to speak and understand Cantonese
* Able to provide informed oral and written consent

Exclusion Criteria:

* Revision total knee replacement
* Single stage bilateral total knee replacement
* Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors
* History of chronic pain other than chronic knee pain
* History of insulin dependent diabetic mellitus, but not diabetic mellitus on oral hyperglycaemic agents
* History of hepatitis B or C carrier
* History of peptic ulcer
* Hx of tuberculosis
* History of immunosuppression
* Daily use of glucocorticoids
* Daily use of strong opioids (morphine, fentanyl, hydromorphone, ketobemidone, methadone, nicomorphine, oxycodone, or meperidine)
* History of severe heart disease (NYHA 2)
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120micromol/L
* Pre-existing neurological or muscular disorders
* Psychiatric illness or neurologic or psychiatric diseases potentially influencing pain perception
* Impaired or retarded mental state
* Difficulties in using patient controlled analgesia (PCA)
* Pregnancy
* Local infection
* On immunosuppresants
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
pain score | at postoperative day 1
  Pain will be measured using numerical rating scale from 0 to 10 with 0 is no pain and 10 is the worst pain

SECONDARY OUTCOMES:
quality of recovery | at postoperative day 1
  quality of recovery will be measured using Quality of Recovery Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wai Cheung, MD, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan TCW, Cheung CW, Wong SSC, Chung AYF, Irwin MG, Chan PK, Fu H, Yan CH, Chiu KY. Preoperative dexamethasone for pain relief after total knee arthroplasty: A randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1157-1167. doi: 10.1097/EJA.0000000000001372. PMID 33105245